CLINICAL TRIAL: NCT01669681
Title: Medical Economic Evaluation of the Care of the Severe Asthma : Cohort COBRA
Brief Title: Cobra (Severe Asthma)Medical-economic
Acronym: Cobra
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8871; 2011-A0156-35 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2012-04-03; First posted 2012-08-21 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Allergic Asthma
Keywords: Severe asthma; Medical economic; care; Cost efficiency; CPAM; EQ5D
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Included in the cohort COBRA

SUMMARY:
The severe asthma is a major source of expenses in term of public health, while it concerns no more than 5 % of the asthmatics. The expenses is direct (medicines, hospitalizations, care) but especially indirect (absenteeisms, etc.). The forward-looking follow-up of cohort of more than 500 severe asthmatic patients multicentrique in an already widely established cohort (COBRA, at present in Visit 9 (one every 6 months) is an once-in-a-lifetime opportunity, coupled with the data of the CPAM, to identify well the evolution in time of a real medical economic variable. The possibility of dynamic follow-up of the expenses compared to the medical data offers perspectives of evaluation cost-efficiency of the informed therapeutic procedures. It is possible to couple in a forward-looking and dynamic way the data of health stemming from a cohort with the economic data stemming from the CPAM. This variable included in a Cluster's algorithm has to allow to identify the interventions the more and the less cost effective. The main objective of this study is to realize a cost estimate of care of the severe asthma. The variation of the costs will be also studied. The recruited patients are patients already included in the cohort COBRA in the centers of Marseille, Montpelier or Nice, classified GINA 4 and agreeing to participate.

DETAILED DESCRIPTION:
The following direct medical costs will be collected according to the point of view of the Social Security on a duration of 2 years:

* Hospitalizations (valuation from the GHS + medicines except GHS)· Consultations (valuation AM)
* Complementary(additional) examinations except hospitalization (valuation AM)
* Pharmacy (valuation AM)
* Transport (valuation AM)The estimate of average costs will be made with a reliable interval for 95 %.

The average cost by patient of the care will be calculated for every year of the follow-up. Relationship individual cost-efficiency: by analogy with the studies cost-efficiency comparative clauses, the investigators shall calculate a relationship cost-efficiency at the individual level as follows: (cost-year2 - cost-year1) / (efficiency-year2 - efficiency-year 1). Differences in these relationships will be looked for between various groups by tests of comparisons of averages.The construction of patients' clusters will be made according to the algorithm of the study SARP but also by using techniques statistics of classification non supervising to define our own algorithm. Variables used on our algorithm will include the relationship cost efficiency individual in addition to the clinical variables. The temporal stability of the relationship cost efficiency will be analyzed. The risk factors of a modification of this relationship will be looked for.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the observationnal cohort COBRA for at least 6 months
* Patient members in one of the partner health insurance funds

Exclusion Criteria:

* The patient refusing his participation to the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruited patients are patients already included in the observationnelle cohort COBRA in the centers of Marseille, Montpelier or Nice, classified GINA 4 and agreeing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
The costs will be updated at the rate recommended by the College of the Economists of the Health. For every year of follow-up will be calculated the individual costs and the annual average cost | Baseline
  The costs will be updated at the rate recommended by the College of the Economists of the Health. For every year of follow-up will be calculated the individual costs and the annual average cost (with a reliable interval in 95 %).

SECONDARY OUTCOMES:
The clinical data will allow to measure the efficiency (control, exacerbation, hospitalization, composite score integrating these various variables). | Baseline
  * The clinical data will allow to measure the efficiency (control, exacerbation, hospitalization, composite score integrating these various variables).
  * The relationship cost efficiency can so be calculated for two years for which we shall have the data.
  * The utility will be measured by means of the validated questionnaire EQ 5D.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOLINARI, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France